CLINICAL TRIAL: NCT04891952
Title: Measuring the Impact of Onco4D® Guidance
Brief Title: Measuring the Impact of Onco4D® Guidance on Chemotherapy Selection and Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Animated Dynamics, Inc. (Industry)
Collaborators: Purdue University (Other)
Responsible Party: Sponsor
Other Study IDs: 003
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Cancer; Chemotherapy Effect
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Onco4D Biodynamic Chemotherapy Selection Assay — Functional precision medicine test to predict response to candidate chemotherapeutic agents

SUMMARY:
Millions of cancer patients each year receive chemotherapy causing adverse side effects that lower quality of life without prolonging it. Reliable identification of ineffective therapies can eliminate needless human suffering while increasing overall probability of positive response to treatment. Chemotherapy resistance profiling entails testing whether a patient exhibits strong resistance to a therapy prior to its final selection by the oncologist.

The Onco4D® chemotherapy selection assay has recently emerged as means to measure the response of intact tumor biopsies to applied therapeutics by using Doppler detection of infrared light scattered from intracellular motions inside living tissue (known as Motility Contrast Tomography or MCT). Several studies have shown this phenotypic profiling technique to offer high accuracy predicting response and resistance to chemotherapy[1-5].

DETAILED DESCRIPTION:
SPECIFIC AIMS The scope of this study is to measure the impact of Onco4D® therapy guidance on treatment and outcomes among cancer patients for whom the test is ordered.

PRIMARY ENDPOINT: Difference in pathologic complete response (pCR) to neoadjuvant chemotherapy among recipients of Onco4D® guided therapy as compared to baseline unguided pCR rates.

SECONDARY ENDPOINTS: Difference in distribution of chemotherapy regimens among recipients of Onco4D® guided therapy as compared to baseline unguided regimens, adjuvant chemotherapy response, 2 and 5 year event free survival (EFS), pre- and post-chemotherapy cancer staging scores (TNM, ACJJ, RCB, etc..), radiologic chemotherapy response, additional exploratory endpoints as appropriate

RESEARCH DESIGN AND METHODS

STUDY DESIGN: Non-randomized multi-center prospective outcomes registry

PARTICIPANT IDENTIFICATION: Cancer patients of all races and ethnic groups are eligible for this registry. All patients treated at participating sites and meeting the inclusion criteria will be offered the opportunity to participate in the registry. Potential participants will be presented with the purpose of the study and the potential risks and benefits of participation. Participants will be considered registered to the study upon receipt of a signed informed consent statement. Registration information will be maintained by the Principal Investigator. All participants will be assigned a unique study ID.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven cancer of any type
2. Onco4D® test ordered by treating physician
3. Ability to understand and willingness to sign an informed consent
4. ≥ 18 years old at time of consent

Exclusion Criteria:

n/a

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients of all races and ethnic groups are eligible for this registry. All patients treated at participating sites and meeting the inclusion criteria will be offered the opportunity to participate in the registry. Potential participants will be presented with the purpose of the study and the potential risks and benefits of participation. Participants will be considered registered to the study upon receipt of a signed informed consent statement. Registration information will be maintained by the Principal Investigator. All participants will be assigned a unique study ID.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2031-08-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) to neoadjuvant chemotherapy | 1 year
  Difference in pathologic complete response (pCR) to neoadjuvant chemotherapy among recipients of Onco4D® guided therapy as compared to baseline unguided pCR rates

SECONDARY OUTCOMES:
Distribution of chemotherapy regimens prescribed | 1 year
  Distribution of chemotherapy regimens prescribed
2 and 5 year Event Free Survival (EFS) | 2 and 5 years
  2 and 5 year Event Free Survival (EFS)
radiologic chemotherapy response | 1 year
  radiologic chemotherapy response

CONTACTS AND LOCATIONS:
Locations (1):
- Animated Dynamics, Inc., Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whitacre E, Manahan E, Burak W, Morgan T, An R, Loesch D: Abstract P3-11-17: A novel biodynamic imaging assay predicts success or failure of neoadjuvant chemotherapy in breast cancer patients. Cancer Research 2019, 79(4 Supplement):P3-11-17.
- [Background] Turek JJ, Nolte DD, An R: Abstract 2849: Biodynamic imaging predicts response of breast cancer patients to neoadjuvant chemotherapy. Cancer Research 2018, 78(13 Supplement):2849.
- [Background] Choi H, Li Z, Sun H, Merrill D, Turek J, Childress M, Nolte D. Biodynamic digital holography of chemoresistance in a pre-clinical trial of canine B-cell lymphoma. Biomed Opt Express. 2018 Apr 17;9(5):2214-2228. doi: 10.1364/BOE.9.002214. eCollection 2018 May 1. PMID 29760982
- [Background] Sun H, Merrill D, An R, Turek J, Matei D, Nolte DD. Biodynamic imaging for phenotypic profiling of three-dimensional tissue culture. J Biomed Opt. 2017 Jan 1;22(1):16007. doi: 10.1117/1.JBO.22.1.016007. PMID 28301634
- [Background] Merrill D, An R, Sun H, Yakubov B, Matei D, Turek J, Nolte D. Intracellular Doppler Signatures of Platinum Sensitivity Captured by Biodynamic Profiling in Ovarian Xenografts. Sci Rep. 2016 Jan 6;6:18821. doi: 10.1038/srep18821. PMID 26732545